CLINICAL TRIAL: NCT04155944
Title: Dr. Pao-Lin Kuo (Department of Obstetrics and Gynecology)
Brief Title: Diagnosis of Prader-Willi Syndrome and Angelman Syndrome
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER-102-155-t
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2018-08

CONDITIONS: Mental Disorder; Fetus Disorder
Keywords: M-PCR; FISH; MLPA; deletion; uniparental disomy; imprinting mutation
MeSH Terms: conditions — Mental Disorders; Fetal Diseases; Uniparental Disomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — fetal DNA extracted from amniocyte, cord blood, or chorionic villus

SUMMARY:
In a retrospective study, data were assessed from cases regarding PWS/AS that underwent molecular diagnosis at the National Chen-Kung University Hospital, Tainan, Taiwan, between January 2001 and December 2014.

DETAILED DESCRIPTION:
Prader-Willi syndrome (PWS) and Angelman syndrome (AS) are two distinct syndromes of developmental impairment that result from loss of the expression of imprinted genes on the q11-q13 region of chromosome 15 (15q11-q13). Approximately 70%--75% of individuals affected with PWS and AS have an interstitial deletion of 15q11-q13. Regarding the remaining individuals with PWS, maternal uniparental disomy is the cause in 20% of cases, imprinting errors in 3% of cases, and chromosomal translocation in approximately 1% of cases. Regarding the remaining cases of AS, paternal uniparental disomy accounts for 2% of cases and mutations in the UBE3A gene for 20% of cases.The PWS/AS critical region was examined by fluorescence in situ hybridization (FISH), methylation-specific PCR (M-PCR), and methylation-specific multiplex-ligation dependent probe amplification(MS-MLPA). In a retrospective study at the National Chen-Kung University Hospital,Tainan, Taiwan, data were reviewed from cases that were referred for molecular diagnosis between January 1, 2001, and December 31, 2014.

ELIGIBILITY:
Inclusion Criteria:

* Individual with clinical features related to Prader-Willi syndrome or Angelman syndrome;
* Fetus with suspicious deletion or duplication of chromosome 15q11.2-q13 visible by the microscope;
* Fetus whose mother or father has chromosomal abnormality involving 15q11.2-q13
* Fetus with mosaic trisomy 15

Exclusion Criteria:

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: During January 1, 2001, and December 31, 2014, cases were referred for molecular diagnosis such as individual with clinical features related to Prader-Willi syndrome or Angelman syndrome ; fetus with deletion or duplication of chromosome 15q11.2-q13 visible by the microscope; fetus whose mother or father has chromosomal abnormality involving 15q11.2-q13 and fetus with mosaic trisomy 15
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
M-PCR(methylation-specific PCR) | up to 4 weeks after diagnosis
  Abnormal pattern of M-PCR can identify PWS or AS
FISH(fluorescent in-situ hybridization) | up to 4 weeks after diagnosis
  A "FISH" test will identify PWS/AS due to a deletion, but it will not identify those by UPD or an imprinting error.
STR(short tandem repeat) for UPD (uniparental disomy) | up to 4 weeks after diagnosis
  A '"STR" test can identify PWS/AS duo to paternal or maternal UPD.
MS-MLPA (methylation-specific multiplex-ligation-dependent probe amplification) | up to 4 weeks after diagnosis
  Use of the quantitative MS-MLPA method provides detailed information about deletions, rare duplications, and possibly UPD

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Lin Kuo, MD, Study Director — Department of Obstetrics and Gynecology, National Chen-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan